CLINICAL TRIAL: NCT02047227
Title: A Phase III, Randomized, Controlled, Single-blind, Multicentre, Parallel Arm Trial to Assess the Efficacy and Safety of Pergoveris® (Follitropin Alfa and Lutropin Alfa) and GONAL-f® (Follitropin Alfa) for Multifollicular Development as Part of an Assisted Reproductive Technology Treatment Cycle in Poor Ovarian Responders, as Defined by the European Society of Human Reproduction and Embryology Criteria
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Pergoveris® in Assisted Reproductive Technology (ESPART)
Acronym: ESPART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR200061-005; 2013-003817-16 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: ESPART; Reproductive Techniques, Assisted; Infertility; Pergoveris®; GONAL-f®
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — pergoveris; follitropin alfa; Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pergoveris® (Experimental)
  Interventions: Drug: Pergoveris®; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- GONAL-f® (Active Comparator)
  Interventions: Drug: GONAL-f®; Drug: Recombinant human chorionic gonadotrophin (r-hCG)

INTERVENTIONS:
Drug: Pergoveris® — Pergoveris (follitropin alfa and lutropin alfa) was administered subcutaneously once daily with a starting dose of 300 International Unit (IU) recombinant human follicular stimulating hormone (rhFSH)/ 150 IU recombinant human luteinizing hormone (rhLH) after confirmation of down regulation up to 21 days. After follicle attained mean diameter of 17-18 millimeter (mm); 250 microgram (mcg) of r-hCG (Ovidrel) was administered once subcutaneously to trigger final follicular maturation as per site standard practice. The dose adjustment for r-hFSH was allowed in 75 IU increments while maintaining the 2:1 ratio of r hFSH to r-hLH in the Pergoveris group based on the subject's response per site standard clinical practice.
  Other Names: r-hFSH/r-hLH; Follitropin alfa/Lutropin alfa
  Arms: Pergoveris®
Drug: GONAL-f® — GONAL-f (r-hFSH) was self-administered subcutaneously once daily at a starting dose of 300 IU after confirmation of down regulation up to 21 days. After follicle attained mean diameter of 17-18 mm; 250 mcg of r-hCG was administered once subcutaneously to trigger final follicular maturation as per site standard practice. The dose adjustment for r-hFSH was allowed in 75 IU increments based on the subject's response per site standard clinical practice.
  Other Names: r-hFSH; Follitropin alfa
  Arms: GONAL-f®
Drug: Recombinant human chorionic gonadotrophin (r-hCG) — On r-hCG day, 250 mcg of r-hCG was administered once subcutaneously
  Other Names: Ovidrel®; Ovitrelle®; choriogonadotropin alfa

SUMMARY:
This is a Phase 3, randomized, controlled, single-blind, multicenter, parallel-arm trial to assess the safety and efficacy of Pergoveris® (recombinant human follicle stimulating hormone [r-hFSH]/recombinant human luteinising hormone [r-hLH]) and GONAL-f® for multifollicular development as part of an assisted reproductive technology (ART) treatment cycle in poor ovarian responders, as aligned with the 2011 Consensus Meeting of the European Society of Human Reproduction and Embryology (ESHRE) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Poor ovarian responders according to specific criteria that are aligned with poor ovarian response (POR) criteria defined by the 2011 Consensus Meeting of the European Society of Human Reproduction and Embryology (ESHRE) as mentioned in the protocol
* Female subjects, less than (<) 41 years of age (according to date of birth at time of informed consent) who are eligible for ovarian stimulation and ART treatment, including intracytoplasmic sperm injection (ICSI)
* Absence of anatomical abnormalities of the reproductive tract that would interfere with implantation or pregnancy
* Absence of any medical condition in which pregnancy is contraindicated
* Body mass index 18 to 30 kilogram per square meter (kg/m^2), inclusive
* Motile, ejaculatory sperm must be available (donated and/or cryopreserved sperm is allowed). Intracytoplasmic sperm injection will be allowed during this trial
* Minimum of 1 month without treatment with either clomiphene citrate or gonadotrophins prior to screening
* Signed and dated informed consent indicating that the subject has been informed of all the pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Two episodes of POR after maximal stimulation
* History or presence of tumors of the hypothalamus or pituitary gland
* History or presence of ovarian enlargement or cyst of unknown etiology, or presence of an ovarian cyst greater than 25 mm on the day of randomization
* Presence of endometriosis Grade III - IV, confirmed or suspected
* Presence of uni- or bilateral hydrosalpinx
* Abnormal gynecological bleeding of undetermined origin
* Contraindication to being pregnant and/or carrying a pregnancy to term
* History or presence of ovarian, uterine or mammary cancer
* Use of testicular or epididymal sperm
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 939 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Result] Humaidan P, Chin W, Rogoff D, D'Hooghe T, Longobardi S, Hubbard J, Schertz J; ESPART Study Investigatorsdouble dagger. Efficacy and safety of follitropin alfa/lutropin alfa in ART: a randomized controlled trial in poor ovarian responders. Hum Reprod. 2017 Mar 1;32(3):544-555. doi: 10.1093/humrep/dew360. PMID 28137754
- [Derived] Humaidan P, Schertz J, Fischer R. Efficacy and Safety of Pergoveris in Assisted Reproductive Technology--ESPART: rationale and design of a randomised controlled trial in poor ovarian responders undergoing IVF/ICSI treatment. BMJ Open. 2015 Jul 3;5(7):e008297. doi: 10.1136/bmjopen-2015-008297. PMID 26141305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 101 sites in 15 countries.
Groups:
- Pergoveris: Pergoveris (follitropin alfa and lutropin alfa) was administered subcutaneously once daily with a starting dose of 300 International Unit (IU) recombinant human follicular stimulating hormone (rhFSH)/ 150 IU recombinant human luteinizing hormone (rhLH) after confirmation of down regulation up to 21 days. After follicle attained mean diameter of 17-18 millimeter (mm); 250 microgram (mcg) of recombinant human chorionic gonadotrophin (r-hCG) (Ovidrel) was administered once subcutaneously to trigger final follicular maturation as per site standard practice. The dose adjustment for r-hFSH was allowed in 75 IU increments while maintaining the 2:1 ratio of r hFSH to r-hLH in the Pergoveris group based on the subject's response per site standard clinical practice.
- GONAL-f: GONAL-f (r-hFSH) was self-administered subcutaneously once daily at a starting dose of 300 IU after confirmation of down regulation up to 21 days. After follicle attained mean diameter of 17-18 mm; 250 mcg of r-hCG was administered once subcutaneously to trigger final follicular maturation as per site standard practice. The dose adjustment for r-hFSH was allowed in 75 IU increments based on the subject's response per site standard clinical practice.
Period: Overall Study
Arm/Group | Pergoveris | GONAL-f
Started | 462 | 477
Completed Ovarian Stimulation Phase | 424 | 440
Completed | 318 | 347
Not Completed | 144 | 130
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Spontaneous pregnancy | 1 | 0
Not completed — Lack of ovarian response to stimulation | 35 | 32
Not completed — No oocytes retrieved | 21 | 20
Not completed — No fertilization | 61 | 51
Not completed — Intention to freeze all embryos | 1 | 0
Not completed — All embryos discarded | 12 | 11
Not completed — Other | 10 | 9

BASELINE CHARACTERISTICS:
Population: All Randomized Subjects Set included all subjects who were randomized.
Groups:
- Pergoveris: Pergoveris (follitropin alfa and lutropin alfa) was administered subcutaneously once daily with a starting dose of 300 IU rhFSH/150 IU rhLH after confirmation of down regulation up to 21 days. After follicle attained mean diameter of 17-18 mm; 250 mcg of r-hCG was administered once subcutaneously to trigger final follicular maturation as per site standard practice. The dose adjustment for r-hFSH was allowed in 75 IU increments while maintaining the 2:1 ratio of r hFSH to r-hLH in the Pergoveris group based on the subject's response per site standard clinical practice.
- Total: Total of all reporting groups
Arm/Group | Pergoveris | GONAL-f | Total
Number analyzed (Participants) | 462 | 477 | 939
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (2.9) | 38.3 (3.0) | 38.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 462 | 477 | 939
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: Mean number of oocytes retrieved on the day of ovum pick up (OPU) was calculated. Oocyte retrieval was a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Time Frame: At approximately 34 to 38 hours after r-hCG administration (Day 113)
Population: Intent-to-treat (ITT) analysis set included all subjects randomized who received at least 1 dose of GONAL-f or Pergoveris.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 462 | 477
oocytes | 3.3 (2.71) | 3.6 (2.82)
Statistical Analysis 1: Comparison: Pergoveris vs GONAL-f; Test type: Superiority or Other; p = 0.054, Poisson Regression Model; Mean Difference (Net) = -0.235, 95% CI 2-sided [-0.4741 to 0.003]

2. Secondary Outcome: Ongoing Pregnancy Rate
Description: Ongoing pregnancy rate was defined as the percentage of subjects with a ultrasound confirmation of at least one viable fetus (positive fetal heart beat).
Time Frame: 70 days after embryo transfer (Day 185)
Population: Modified intent-to-treat (MITT) analysis set included all randomized subjects who received at least 1 dose of GONAL-f or Pergoveris and did not have spontaneous pregnancy or death at approximately 34-38 hours after rhCG administration.
Measure: Number; unit: percentage of subjects
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 462 | 477
percentage of subjects | 11.0 | 12.4

3. Secondary Outcome: Live Birth Rate
Description: Live birth rate was defined as the percentage of subjects with at least one live-born neonate.
Time Frame: Approximately 180 days following ongoing pregnancy determination (Day 365)
Population: MITT analysis set included all randomized subjects who received at least 1 dose of GONAL-f or Pergoveris and did not have spontaneous pregnancy or death at approximately 34-38 hours after rhCG administration.
Measure: Number; unit: percentage of subjects
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 462 | 477
percentage of subjects | 10.6 | 11.7

4. Secondary Outcome: Embryo Implantation Rate
Description: Embryo implantation rate was measured as the number of gestational sacs observed divided by the number of embryos transferred multiplied by 100.
Time Frame: 35-42 days post r-hCG administration (Day 154)
Population: MITT analysis set included all randomized subjects who received at least 1 dose of GONAL-f or Pergoveris and did not have spontaneous pregnancy or death at approximately 34-38 hours after rhCG administration. Here "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: percent sacs per embryo
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 319 | 349
percent sacs per embryo | 14.7 | 15.6

5. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy rate defined as the percentage of subjects with a ultrasound confirmation of a gestational sac, with or without fetal heart activity.
Time Frame: 35-42 days post r-hCG administration (Day 154)
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 462 | 477
percentage of subjects | 14.1 | 16.8

6. Secondary Outcome: Biochemical Pregnancy Rate
Description: Biochemical pregnancy rate was defined as the percentage of subjects with a positive beta-hCG result from the serum pregnancy test.
Time Frame: 15 to 20 days post r-hCG administration (Day 132)
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Pergoveris | GONAL-f
Number analyzed (Participants) | 462 | 477
percentage of subjects | 17.3 | 23.9

ADVERSE EVENTS:
Time Frame: Baseline up to 180 days after ongoing pregnancy (maximum up to 365 days)
Arm/Group | Pergoveris | GONAL-f
Serious Adverse Events (participants affected / at risk) | 8/462 | 17/477
Other Adverse Events (participants affected / at risk) | 111/462 | 151/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pergoveris (N=462) | GONAL-f (N=477)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 | 0
Ovarian rupture (Reproductive system and breast disorders) | 1 | 0
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 | 1
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pergoveris (N=462) | GONAL-f (N=477)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Ear swelling (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 12
Abdominal pain (Gastrointestinal disorders) | 12 | 13
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Abdominal pain lower (Gastrointestinal disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 7
Constipation (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 4
Injection site erythema (General disorders) | 4 | 4
Crying (General disorders) | 2 | 3
Asthenia (General disorders) | 2 | 1
Chest discomfort (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Food allergy (Immune system disorders) | 2 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 2 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 3
Cystitis (Infections and infestations) | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 1 | 2
Sinusitis bacterial (Infections and infestations) | 0 | 2
Bacterial disease carrier (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Body temperature increased (Investigations) | 1 | 4
Weight increased (Investigations) | 1 | 2
Menstruation normal (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Nitrite urine present (Investigations) | 1 | 0
Urine ketone body (Investigations) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 46 | 58
Dizziness (Nervous system disorders) | 4 | 8
Migraine (Nervous system disorders) | 5 | 2
Somnolence (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 2
Head discomfort (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 6 | 12
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 5 | 5
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 3
Mood swings (Psychiatric disorders) | 3 | 1
Nervousness (Psychiatric disorders) | 2 | 2
Agitation (Psychiatric disorders) | 2 | 0
Depressive symptom (Psychiatric disorders) | 1 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Libido increased (Psychiatric disorders) | 1 | 0
Tearfulness (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 2
Leukocyturia (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 6 | 6
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 6
Breast tenderness (Reproductive system and breast disorders) | 3 | 2
Adnexa uteri pain (Reproductive system and breast disorders) | 2 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Nipple disorder (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Premenstrual pain (Reproductive system and breast disorders) | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
Hot flush (Vascular disorders) | 19 | 10
Flushing (Vascular disorders) | 3 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Breast pain (Reproductive system and breast disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No